CLINICAL TRIAL: NCT03680794
Title: sCD160 in Sera and Intra-ocular Fluids: Association With Ischaemic Retinopathies
Brief Title: Soluble Cluster of Differentiation 160 (sCD160) in Sera and Intra-ocular Fluids: Association With Ischaemic Retinopathies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PA18053
Record Dates: First submitted 2018-05-15; First posted 2018-09-21 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Retinopathy; Retinal Vein Occlusion
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with ophthalmic surgery (Experimental)
  Interventions: Other: sampling of ophthalmic liquid

INTERVENTIONS:
Other: sampling of ophthalmic liquid — aqueous sampling for patients with cataract surgery or vitreous sampling for patients with posterior segment surgery

SUMMARY:
CD160 represents a new angiogenic factor as its specific engagement by an agonist monoclonal antibody directed against human CD160 reduced angiogenesis of endothelial cells with a distinct mechanism from current angiogenic therapies that target the VEGF/VEGF-R pathway. A soluble form of CD160, sCD160, has been found to be highly expressed in the vitreous and the sera of patients with severe diabetic retinopathies, and can now be dosed with help of an ELISA test.

The investigators aim to evaluate the association between ischaemic retinopathies (patients with or without) and sCD160 concentrations in the vitreous, the aqueous humour and the serum.

DETAILED DESCRIPTION:
120 patients enrolled for ophthalmic surgery (cataract or posterior segment surgery (epiretinal membrane, macular hole, vitrectomy)) will be recruited in the Department of Ophthalmology, Robert Debré Hospital, Reims, France.

Each patient will benefit a complete ophthalmologic examination, and either an aqueous sampling (cataract) or a vitreous sampling (posterior segment) along with a serum sampling at the beginning of the surgery. ELISA test will be performed on vitreous or aqueous samples in triplicates. Luminex will be performed on vitreous samples in order to determine the concentrations of several ischemia biomarkers (VEGF, PlGF, Platelet-derived growth factor (PDGF-B), SDF-1, Angpt2, InterIeukin IL-6, IL-8, CD105, Monocyte chemoattractant protein 1 (MCP-1), IL-10, interferon-inducible protein-10 ( IP-10), IL-1B and CD106, RAGE).

Primary objective is:

- Evaluation of the association between ischaemic retinopathies (patients with or without) and sCD160 concentrations of the vitreous or the aqueous humours.

Secondary objectives are:

* Evaluation of the association between diabetic retinopathies (patients with or without) and sCD160 concentrations of the vitreous, the aqueous humours and the sera.
* Evaluation of the association between several vitreous biomarkers of ischaemia and sCD160 concentrations of the vitreous and the sera.
* Evaluation of the association between sCD160 concentrations in the vitreous and the sera.
* Evaluation of the association between sCD160 concentration in the aqueous humours and the sera.

ELIGIBILITY:
inclusion criteria :

* over 18 years old
* with social security affiliation
* willing to participate this study non-inclusion criteria :
* any prior (3 months) or concomitant treatment with anti-VEGF therapy, corticosteroids, or immunosuppressive agents
* any history of previous vitreoretinal surgery, ocular tumor, severe ocular trauma, severe intraocular, periocular infection, inflammation, or radiation
* any serious allergy to the fluorescein sodium for injection in angiography
* any history of previous systemic anti-VEGF treatment
* any history of inflammatory or auto-immune disease
* any active extraocular inflammation or infection in the last 4 weeks before surgery exclusion criteria :
* Patients with C-reactive protein CRP > 10mg/mL (serum sampling during surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-06-27 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
sCD160 concentration in the vitreous humor | Day 0
  ELISA test
sCD160 concentration in the aqueous humor | Day 0
  ELISA test

SECONDARY OUTCOMES:
sCD160 concentration in the serum | Day 0
  ELISA test
Diabetic retinopathy severity | Day 0
  Angiography
Vascular endothelial growth factor (VEGF) | Day 0
  LUMINEX test
Placenta Growth Factor-1(PlGF) | Day 0
  LUMINEX test
Stromal cell-derived factor 1 (SDF-1) | Day 0
  LUMINEX test

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided